CLINICAL TRIAL: NCT04555460
Title: Hemicraniectomy in Patients With Malign Middle Cerebral Artery Infarction: A Randomized, Controlled Study
Brief Title: Hemicraniectomy in Patients With Malign Middle Cerebral Artery Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Emre Kumral, Prof. MD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003/44
Record Dates: First submitted 2020-09-08; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Herniation
Keywords: infarction, hemicraniectomy
MeSH Terms: conditions — Infarction | interventions — Decompression, Surgical; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive surgery (Active Comparator): Decompressive surgery was performed with a large hemicraniectomy that removed, ipsilateral to the stroke, a bone flap as large as possible including temporal, frontal, parietal, and some occipital squama.
  Interventions: Procedure: Hemicraniectomy
- Conservative medical therapy (Active Comparator): Conservative medical therapy was based on published guidelines for the early management of patients with ischemic stroke. Administration of intravenous mannitol (0.25 to 0.5 g/kg) or furosemide was given only in patients whose condition was rapidly worsening because of brain edema, without additional recommendations on loading doses.
  Interventions: Other: Conservative medical therapy

INTERVENTIONS:
Procedure: Hemicraniectomy — Large hemicraniectomy and duraplasty
  Other Names: Surgical decompression
  Arms: Decompressive surgery
Other: Conservative medical therapy — Conservative medical therapy was based on published guidelines for the early management of patients with ischemic stroke
  Other Names: Control group
  Arms: Conservative medical therapy

SUMMARY:
This trial is a prospective, randomized, controlled, clinical trial based on a stroke center. We randomly assigned 151 patients 41 years of age or older (median, 65 years; range, 41 to 83) with malignant middle cerebral artery infarction to either conservative medical treatment or hemicraniectomy; assignments were made within 12 to 38 hours after the onset of symptoms. The primary end point was survival with slight or moderate disability 12 months after randomization (defined by a score of 0 to 3 on the modified Rankin scale, which ranges from 0 [no symptoms] to 6 [death]). Secondary outcome included death, Barthel Index, National Institute of Health Stroke Scale, and Stroke Impact Scale 2.0 (SIS) 6 months and 1 year after randomization. Variables for subgroup analyses were age, sex, presence of aphasia or neglect, stroke severity and time to randomization. The study was performed according to Consolidated Standards of Reporting Trials (CONSORT).

DETAILED DESCRIPTION:
Patients between 40 to 80 years of age were included within 12 to 38 hours of a malignant middle cerebral artery infarction defined by the association of 3 criteria: a National Institutes of Health Stroke Scale score ≥16, including a score ≥1 for item 1a (level of consciousness); brain computed tomography ischemic signs involving 2/3 of the middle cerebral artery territory; and a diffusion-weighted imaging (DWI) infarct volume >150cm3. The first patient was enrolled in January 2003 and the last patient in December 2007. An independent data safety monitoring committee monitored the safety, progress, and ethics of the trial. Patients were randomized to either surgical plus medical treatment or to conservative medical treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* A National Institutes of Health Stroke Scale score ≥16
* A score ≥1 for item 1a (level of consciousness)
* Brain computed tomography ischemic signs involving 2/3 of the middle cerebral artery territory
* Diffusion-weighted imaging infarct volume >150cm3

Exclusion Criteria:

* Prestroke modified Rankin score score ≥2
* Prestroke score on the Barthel Index <95
* Score on the Glasgow Coma Scale <6
* Both pupils fixed and dilated
* Any other coincidental brain lesion that might affect outcome
* Plasminogen activator in the 12 h before randomisation
* Space-occupying hemorrhagic transformation of the infarct
* Pregnancy
* Life expectancy <3 years
* Other serious illness that might affect outcome
* Known coagulopathy or systemic bleeding disorder
* Contraindication for anesthesia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-01-23 (Actual); Primary Completion 2007-12-30 (Actual); Study Completion 2008-12-30 (Actual)

PRIMARY OUTCOMES:
modified Rankin score 0-3 | 1 year
  Slight or moderate disability 12 months after randomization (defined by a score of 0 to 3 on the modified Rankin scale

SECONDARY OUTCOMES:
Death | 1 year
  Death at 6 month and 1 year
Barthel Index | 1 year
  measured12 months after randomization (defined by a score of 0 to 100; as 100 being the best)
National Institute of Health Stroke Scale (NIHSS) | 1 year
  measured12 months after randomization (The maximum possible score is 42, with the minimum score being a 0)
Stroke Impact Scale 2.0 (SIS) | 1 year
  The score of each domain was calculated as 100 being the best, with a range of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Timur Köse, PhD, Principal Investigator — Biostatistic Department, Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
3 months after publication data will be shared